CLINICAL TRIAL: NCT01541605
Title: International Randomised Double-blind Placebo-controlled Study on the Initial Treatment of Acute Mania With Methylphenidate
Brief Title: Methylphenidate for the Treatment of Acute Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Michael Kluge (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor-Investigator, Michael Kluge, Senior Psychiatrist, University of Leipzig
Organization: University of Leipzig (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEMAP1
Record Dates: First submitted 2012-02-16; First posted 2012-03-01 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Mania
MeSH Terms: conditions — Mania | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylphenidate (Active Comparator)
  Interventions: Drug: methylphenidate
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate — tablets for oral use
  Arms: methylphenidate
Drug: Placebo — tablets for oral use
  Arms: placebo

SUMMARY:
This study aims at evaluating the efficacy and safety of methylphenidate in the initial treatment of acute mania in patients with bipolar affective disorders.

DETAILED DESCRIPTION:
Mania can be regarded as an autoregulatory mechanism to enhance unstable vigilance. There is increasing evidence that psychostimulants that increase vigilance may be effective in treating mania. However, controlled studies are lacking.

This is a two-arm, randomised, placebo-controlled, double-blind, parallel, multi-centre phase IIIb exploratory study to evaluate the efficacy and safety of methylphenidate in the initial treatment of acute mania in patients with bipolar affective disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients
2. Written informed consent by patients who are competent to consent to study participation.
3. Diagnosis: manic episode according to the International Classification of Diseases 10th Revision (ICD-10): F30.0, F30.1, F31.0 or F31.1
4. Male or female of at least 18 years of age
5. YMRS total score ≥ 20 and ≤ 45 points
6. Body mass index (BMI) > 17
7. Patients must be able to swallow tablets (study drug).

Exclusion Criteria:

1. Any other current major psychiatric ICD-10 disorder is an exclusion criterion except for the following F90, F17.1, F17.2, F40-F59, F60-F69
2. Contraindications for treatment with methylphenidate except as noted otherwise
3. Serious non-psychiatric disease, that may interfere with the objectives of the study or with the safety or compliance of the subject, as judged by the investigator
4. Oral administration of monoaminooxidase (MAO)-inhibitors within two weeks, fluoxetine within 6 weeks and of any other antidepressant or primarily psychotropic substance except for those specified below within one week before study entry.
5. Stable treatment with mood stabilisers including lithium, anticonvulsants (e.g. valproate, carbamazepine) or antipsychotics (e.g. risperidone, olanzapine) or benzodiazepines is NOT an exclusion criterion and will be continued; however, patients receiving more than 2 of these substances are NOT eligible for inclusion
6. Medical history of other disorders of CNS including tics or dyskinesia
7. Medical history of cardiovascular diseases, severe hypertension, glaucoma, hyperfunction of the thyroid
8. Patients with congenital or acquired long QT syndrome, or with a familiy history of QT prolongation, sudden cardiac death or other significant inherited cardiac disorders (e.g. family history of hypertrophic cardiomyopathy).
9. History of Electroconvulsive therapy within the last 3 month
10. Known alcohol and drug addiction or abuse, except for patients with abstinence > 3 month. Patients with sporadic abuse of cannabis (products) will not be excluded from the study. That is even true with a positive Tetrahydrocannabinol (THC) screen in urine.
11. Pregnant or nursing woman
12. Concomitant participation in other clinical trials or participation during the 30 days prior to screening
13. Prior participation in this study
14. Suicidality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
manic symptoms as assessed by the Young Mania Rating Scale (YMRS) | after 2.5 days of treatment

SECONDARY OUTCOMES:
EEG-vigilance as assessed by the Vigilanz Algorhithm Leipzig (VIGALL) | after 2.5 days of treatment
movements as assessed by actimetry | after 2.5 days of treatment
cognitive performance as assesd with the Screen for Cognitive Impairment in Psychiatry (SCIP) | after 2.5 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Hegerl, Prof. Dr., Principal Investigator — University of Leipzig
Locations (10):
- Katholieke Universiteit Leuven, campus Kortenberg, Kortenberg, Belgium
- Germany (4):
  - Universität Bochum, Bochum
  - Universität Dresden, Dresden
  - Universität Halle, Halle
  - Universität Leipzig, Leipzig
- Semmelweis University, Budapest, Hungary
- Spain (4):
  - Hospital Sant Pau, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Universitario la Princesa, Madrid
  - Hospital Santiago Apóstol, Vitoria-Gasteiz

REFERENCES:
- [Background] Kluge M, Hegerl U, Sander C, Dietzel J, Mergl R, Bitter I, Demyttenaere K, Gusmao R, Gonzalez-Pinto A, Perez-Sola V, Vieta E, Juckel G, Zimmermann US, Bauer M, Sienaert P, Quintao S, Edel MA, Bolyos C, Ayuso-Mateos JL, Lopez-Garcia P. Methylphenidate in mania project (MEMAP): study protocol of an international randomised double-blind placebo-controlled study on the initial treatment of acute mania with methylphenidate. BMC Psychiatry. 2013 Feb 27;13:71. doi: 10.1186/1471-244X-13-71. PMID 23446109
- [Derived] Hegerl U, Mergl R, Sander C, Dietzel J, Bitter I, Demyttenaere K, Gusmao R, Gonzalez-Pinto A, Zorrilla I, Alocen AG, Sola VP, Vieta E, Juckel G, Zimmermann US, Bauer M, Sienaert P, Quintao S, Edel MA, Bolyos C, Ayuso-Mateos JL, Lopez-Garcia P, Kluge M. A multi-centre, randomised, double-blind, placebo-controlled clinical trial of methylphenidate in the initial treatment of acute mania (MEMAP study). Eur Neuropsychopharmacol. 2018 Jan;28(1):185-194. doi: 10.1016/j.euroneuro.2017.11.003. Epub 2017 Nov 23. PMID 29174864